CLINICAL TRIAL: NCT03177382
Title: Total Neoadjuvant Treatment Versus Conventional Neo-chemoradiotherapy in Locally Advanced Rectal Cancer With High Risk Factors: a Multicenter Randomized Phase III Clinical Study.
Brief Title: Total Neoadjuvant Treatment vs. Chemoradiotherapy in Local Advanced Rectal Cancer With High Risk Factors
Acronym: TNTCRT
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Ziqiang Wang,MD, Professor, West China Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TNT-2
Record Dates: First submitted 2017-05-31; First posted 2017-06-06 (Actual); Last update posted 2018-05-08 (Actual); Status verified 2018-05

CONDITIONS: Total Neoadjuvant Treatment; Chemoradiotherapy; Local Advanced Rectal Cancer; High Risk Factors
Keywords: Total Neoadjuvant Treatment; Rectal Cancer; High Risk Factors; Chemoradiotherapy
MeSH Terms: conditions — Rectal Neoplasms | interventions — Trinitrotoluene; Chemoradiotherapy; Chemotherapy, Adjuvant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Total neoadjuvant treatment (Experimental): The interventions of experimental group include 1 cycle of CAPOX before radiotherapy; and then start concurrent chemoradiotherapy with CAPOX regimen (capecitabine: 825mg/m2, bid, 5d/w; oxaliplatin, 130mg/m2, D1, q3w) for 2 cycles followed by 3 cycles of CAPOX 2-3 weeks after the completion of radiotherapy. Intensity modulated radiotherapy (IMRT/VMAT) was used for radiotherapy, and the dose was 50-50.4Gy/25-28f, 1.8-2.0Gy/d, 5f/w. The TME operation will be given 3-4 weeks after the end of the total neoadjuvant treatment.
  Interventions: Radiation: Total neoadjuvant treatment; Procedure: TME
- concurrent chemoradiotherapy group (Active Comparator): The interventions of control group is standard preoperative concurrent chemoradiotherapy. The radiotherapy target areas and dosage are the same as group TNT. During radiotherapy, only oral capecitabine will be delivered and capecitabine dose was 825mg/m2, bid, 5d/w. The TME surgery will be performed 6-8 weeks after the end of concurrent chemoradiotherapy. Then, patients will receive another 6 cycles of CAPOX.
  Interventions: Radiation: concurrent chemoradiotherapy; Procedure: TME; Drug: Adjuvant chemotherapy

INTERVENTIONS:
Radiation: Total neoadjuvant treatment — The interventions of experimental group include 1 cycle of CAPOX before radiotherapy; and then start concurrent chemoradiotherapy with CAPOX regimen (capecitabine: 825mg/m2, bid, 5d/w; oxaliplatin, 130mg/m2, D1, q3w) for 2 cycles followed by 3 cycles of CAPOX 2-3 weeks after the completion of radiotherapy. Intensity modulated radiotherapy (IMRT/VMAT) was used for radiotherapy, and the dose was 50-50.4Gy/25-28f, 1.8-2.0Gy/d, 5f/w.
  Other Names: TNT
  Arms: Total neoadjuvant treatment
Radiation: concurrent chemoradiotherapy — The interventions of control group is standard preoperative concurrent chemoradiotherapy. The radiotherapy target areas and dosage are the same as group TNT. During radiotherapy, only oral capecitabine will be delivered and capecitabine dose was 825mg/m2, bid, 5d/w. The TME surgery will be performed 6-8 weeks after the end of concurrent chemoradiotherapy. Then, patients will receive another 6 cycles of CAPOX.
  Other Names: CRT
  Arms: concurrent chemoradiotherapy group
Procedure: TME — The TME operation will be given after the end of the neoadjuvant treatment.
Drug: Adjuvant chemotherapy — Patients will receive another 6 cycles of CAPOX after TME.
  Arms: concurrent chemoradiotherapy group

SUMMARY:
Purpose:To compare the efficacy and the safety of total neoadjuvant chemotherapy + TME with standard neoadjuvant concurrent chemoradiotherapy + TME + adjuvant chemotherapy for locally advanced rectal cancer patients with high risk factors of recurrence.

Evaluation indexes: (1) the primary evaluation index: disease-free survival (disease free survival, DFS); (2) the secondary evaluation indexes: pathological complete remission rate (pCR), the 3 year overall survival (overall survival, OS); R0 dissection rate; distant metastasis free survival (DMFS); local recurrence free survival rate (LRRFS); tumor regression grade (TRG, tumor regression grade) and the adverse reaction rate during the chemotherapy, the operation safety index; quality of life; psychological and cognitive effects, assessment of nutritional status.

Safety evaluation indexes: including all adverse events observed during the experiment.

Number of patients: 458 cases Study design: patients will be randomly assigned into the total neoadjuvant treatment group (experimental group, TNT) and neoadjuvant concurrent chemotherapy group (control group, CRT) in the ratio of 1: 1. The patients of experimental group will be given 1 cycle of induction CAPOX (Oxaliplatin 130mg/m2 d1, Capecitabine 1000mg/m2, bid, d1-14) prior to radiotherapy. Then pelvic IMRT/VMAT (50-50.4Gy/25-28f) and two cycles of concurrent chemotherapy (Oxaliplatin 130mg/m2, d1, d 22, Capecitabine 825mg/m2, bid, 5d/w, 25-28d) are performed. And three cycles of consolidation chemotherapy (CAPOX) are delivered after concurrent chemoradiotherapy. Total mesorectal excision (TME) is performed after completion of the whole neoadjuvant treatment. The patients of control group will receive standard concurrent neoadjuvant chemoradiotherapy with capecitabine (825mg/m2, bid, 5d/w) followed by TME 6-8 weeks after the end of concurrent chemoradiotherapy. Then, patients are treated with another 6 cycles of CAPOX.

Schedule: Investigators plan to finish the study in 4 years and write the related work within 2 years after the completion of this study.

ELIGIBILITY:
Inclusion Criteria:（1）Age: 18 ~ 70 years old; sex is not limited. （2）Patients with stage II/III rectal cancer staged under MRI or endoscopic ultrasonography and have at least one risk factor: cT4a-b(resectable)；cT3c-d with EMVI+ (Extramural venous invasion)；cN2；MRF+ (MRI in evaluating the mesorectal fascia).（According to the 2010 AJCC cancer staging system, the seventh edition）. The preoperative T stage is referred to endoscopic ultrasonography or rectal MRI. The N stage is referred to abdominal CT. The M stage is referred to abdominal and thoracic CT. If symptoms occur, other appropriate imaging examinations are needed（cranial MRI or ECT）.

（3）The lower edge of lesion is less than 12cm from anal verge according to rigid sigmoidoscopy or rectal digital examination.

（4）No distant metastasis after a thorough examination . （5）Pathological diagnosis of rectal adenocarcinoma. （6）ECOG score: 0-1. （7）Patients with primary rectal cancer who had not received surgery prior to surgery (except for palliative ileostomy or colostomy), radiotherapy, systemic chemotherapy or other anti-tumor therapy.

（8）The main organ function is normal, including the following characteristics:

* Blood routine examination: HB ≥9g/dL, WBC ≥ 3.5/4.0×109/L，PLT≥ 100×109/L

  * Biochemical examination：Crea and BIL ≤ 1.0 upper normal limit（ULN），ALT and AST≤ 2.5 upper normal limit（ULN）.

    （9）Not allergic to 5-Fu or Platinum. （10）The site of radiotherapy had not previously received radiation. （11）If female and of childbearing potential, have a negative result on a pregnancy test performed a maximum of 7 days before initiation of study treatment. If female and of childbearing potential, or if male, agree to use adequate contraception (eg, abstinence, intrauterine device, oral contraceptive, or double-barrier method) based on the judgment of the investigator or a designated associate from the date on which the ICF (Informed Consent Form) is signed until 8 weeks after the last dose of study drug.

    （12）Participants are volunteered to participate in this study, sign informed consent, good compliance, cooperation with follow-up.

Exclusion Criteria:（1）Have had prior or concurrent cancer distinct in primary site or histology EXCEPT for curatively treated cervical cancer in situ, Basal cell carcinoma of skin.

（2）Pregnant or lactating women. （3）Patients with severe cardiovascular disease and poorly controlled diabetes. （4）Mental disorder. （5）Severe infection. （6）Patients who can't finish MRI examination. （7）Patients were treated with thrombolytic therapy and anticoagulant therapy, either with bleeding diathesis or coagulopathy, or aneurysm, stroke, transient ischemic attack, arteriovenous malformation in the past year.

（8）The past history of kidney disease, urine or urine protein found in clinical renal abnormalities.

（9）The digestive tract fistula, perforation or serious ulcer disease. （10）Be allergic to 5-Fu or Platinum. （11）The presence of severe gastrointestinal diseases that affecting the absorption of oral chemotherapy drugs.

（12）Additional clinical trials were attended within 4 weeks before treatment initiation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 458 (Estimated)
Dates: Start 2017-06-15 (Actual); Primary Completion 2021-05-30 (Estimated); Study Completion 2023-05-30 (Estimated)

PRIMARY OUTCOMES:
disease free survival | 3 years
  Time from the completion of the treatment to any recurrences or distant metastases

SECONDARY OUTCOMES:
pathological complete remission rate | 1 months
  The rate of complete remission patients to all resected patients
the 3 year overall survival rate | 3 years
  The rate of patients alive 3 years after the completion of treatment
R0 dissection rate | 1 months
  The rate of patients who received R0 dissection to all the patients
distant metastasis free survival | 3 years
  Time from the completion of the treatment to any distant metastases
local recurrence free survival rate | 3 years
  The rate of patients without local recurrence to all the patients
tumor regression grade (TRG) | 1 months
  The level of tumor regression under pathological examination
the adverse effects during the chemotherapy | 3 months
  Any side effects during the chemotherapy
the operation safety index | 3 months
  The safety index of operation
quality of life | 3 years
  Patients' subjective feeling of life
psychological and cognitive effects | 3 years
  The psychological and cognitive changes of patients after treatment
assessment of nutritional status | 6 months
  The nutritional status of patients

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - West China Hospital, Chengdu, Sichuan
  - The Second Affiliated Hospital of Zhejiang University, Hanzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No